CLINICAL TRIAL: NCT05446064
Title: Buddhism Beliefs and HIV Stigma in Thailand: An Intervention Study
Brief Title: Buddhism Beliefs and HIV Stigma in Thailand
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The NIH terminated the award prematurely.
Sponsor: University of California, Los Angeles (Other)
Collaborators: Chiangmai Rajabhat University (Unknown)
Responsible Party: Principal Investigator, Weiti Chen, RN, CNM, PhD, FAAN, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB#22-000560
Record Dates: First submitted 2022-06-24; First posted 2022-07-06 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections; Stigma, Social; Care Eliciting Behavior
Keywords: People living with HIV; Stigma; Buddhism; Intervention testing
MeSH Terms: conditions — HIV Infections; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Treatment (Experimental): Participants will receive the stigma-reduction intervention as well as typical services including care co-ordination and linkage to public health nurses in local communities.
  Interventions: Behavioral: Stigma-reduction intervention
- Treatment-as-Usual (No Intervention): Participants will receive typical services including care co-ordination and linkage to public health nurses in local communities.

INTERVENTIONS:
Behavioral: Stigma-reduction intervention — The intervention is modularized into four weekly 1-hour group sessions, led by a trained facilitator who provides psychoeducation to promote awareness and understanding of HIV stigma and teach CBT-based coping skills. Each group session will last 45-60 minutes. Participants are introduced to the general CBT model of HIV stigma and encouraged to track thoughts, feelings, and behavioral responses when encountering external stigma or adverse events. The participants further learn to differentiate effective and ineffective coping strategies and practice applying new coping skills to reduce internalized HIV stigma. The interventionist will follow the intervention manual to deliver the intervention and assign homework for group members to practice on their own. In the following sessions, the interventionist will review progress with participants, guide participants through exercises, and identify additional problems to be addressed in subsequent sessions.
  Arms: Enhanced Treatment

SUMMARY:
Thailand remains one of the countries with the largest population of people living with HIV (PLWH). It is estimated that 30 Thai provinces account for 75% of the HIV infections in that country, with ChiangMai as the most prevalent province in northern Thailand. Also, HIV/AIDS remains among the top 10 most common causes of death in Thailand. This high mortality rate may be partially explained by the notable HIV treatment cascade in Thailand: Among all the Thai PLWH, only 74% were retained in care, while 68% received ART, and roughly 50% reached viral suppression. An important reason for this is that HIV-related stigma still poses significant barriers for Thai PLWH to access healthcare and carry out health-protective behaviors, including adherence to medication schedules, to manage their HIV. In Thailand, substance use, including use of tobacco, alcohol, and other emerging recreational drugs, is a pressing health concern. In the HIV+ population in Thailand, it was found that 15% use tobacco, 70% use alcohol, and 2% use recreational drugs. In addition, among Thai HIV+ alcohol drinkers, about 13%-22% were heavy drinkers and 40% had sex under the influence of alcohol. Although the literature evaluating prevalence of substance use among Thai HIV+ individuals is emerging, the knowledge remains very limited regarding their risk and protective factors for substance use. Self-management interventions, typically include training modules for symptom management skills and coping strategies. In Buddhist-Thai culture, the goal of self-management may become assisting PLWH to find the peace and harmony within themselves by gradually "letting go" of those strong desires for certain materials or status that contribute to the uncertainty in lives. Therefore, this project aims to further the investigator's knowledge about self-management behaviors in HIV+ substance users in the context of Buddhist-Thai culture. The investigator aims to: 1. Explore how PLWH experience and interpret substance use, mental health, and self-management and identify key social-cultural factors that influence these factors. 2. Test the associations among mental health, substance use, self-management, health outcomes and selected key social-cultural factors among PLWH using a partial correlation network model. The results will be used for development of a culturally tailored, evidence-based self-management intervention to promote better health outcomes among Thai PLWH.

DETAILED DESCRIPTION:
HIV Stigma and Health among People Living with HIV (PLWH):

Stigma is a primary risk factor affecting the well-being and survival of PLWH, in particular PLWH who are marginalized by society. HIV has long been a highly stigmatized disease, and researchers have made great efforts to study various dimensions of HIV stigma, resulting in an established body of literature. HIV stigma is conceptualized as "a collection of adverse attitudes, beliefs, and actions" of others against PLWH (external stigma), which may result in "internalized beliefs or actions" taken by PLWH (internal stigma), leading to negative health outcomes. Three decades of research have converged, demonstrating that HIV stigma, both external and internal, can negatively impact the well-being and survival of PLWH across the globe through multiple pathways. Populations that have been socially marginalized, such as women, ethnic minorities, and sexual and gender minorities, are particularly vulnerable to the negative impact of HIV stigma. HIV stigma is a huge barrier to accessing social support and health services, with negative impacts on PLWH's mental health and optimal self-management of their HIV, such as adherence to medication. For PLWH in Asia, HIV stigma negatively impacts mental health and HIV self-managing behaviors, leading to deteriorated subjective well-being, physical health, and survival.

HIV Epidemic and AIDS Care System in Thailand:

Thailand has the highest HIV prevalence rate in the Asian-Pacific region, with an estimated 1.2% of its adult population infected. Because of this high prevalence rate, Thailand remains one of the countries with the largest number of people living with HIV (PLWH) in the Asia-Pacific region. Thailand only follows India, China, and Indonesia in number of PLWH, although its population size is ranked 11th in the region. Currently there are 0.5 million PLWH living in Thailand. Although, historically, HIV affected mostly female sex workers and their clients in Thailand, the HIV epidemic has changed drastically due to proactive interventions in the 1990s. Recently, the HIV epidemic has come to resemble those in other developed countries, with men who have sex with men (MSM; 9.2-40%), transgender individuals (12%), sex workers (1-16%), and substance users (19%) sharing the increasing burdens of HIV. Additionally, due to unequal distributions of vulnerable populations and risk factors for HIV infection, it is estimated that 30 Thai provinces account for 75% of the country's HIV infections, with Chiang Mai being one of the provinces having the highest prevalence.

As part of its response to the HIV epidemic, the Thai government began to provide free antiretroviral treatment (ART) for PLWH with impaired immune functions (≤ CD4 350 cell/mm3) in the early 2000s. It then expanded the program to all PLWH, regardless of their immune function, in 2014. This policy has enabled high ART accessibility in Thailand, making it one of the few countries in Asia-Pacific region that has more than 50% of PLWH to be on ART. Due to high ART coverage, Thailand experienced success in reducing HIV mortality: an estimated 196,000 deaths were averted between 2001 and 2014. In addition, Thai PLWH increased their life expectancy to 71 years old or longer, which is close to that of the general Thai population. Despite these important gains, however, the number of PLWH has constantly decreased by approximately 10,000 per year over the past decade, which could be attributed to high mortality rates that surpassed incidence rates. In 2016, it was estimated that while there were 6,400 new HIV cases, there were 16,000 HIV-related deaths, resulting in an overall mortality rate of 3.56%. Compared with the 0.6% mortality rate in the United States during the same period, the mortality rate in Thailand remained 5 times higher. Indeed, HIV still remains one of the top 10 most common causes of death in Thailand. This high mortality rate may be partially explained by the notable HIV treatment cascade in Thailand: among all Thai PLWH, 74% were retained in care, 68% received ART, and only roughly 50% reached viral suppression. An important reason for the low viral suppression rate is that HIV remains a highly stigmatized disease in Thailand, HIV-related stigma still poses significant barriers for Thai PLWH to access healthcare and carry out health-protective behaviors to manage their HIV, including adherence to medications.

HIV Stigma among People Living with HIV in Thailand:

As Thailand was one of the early epicenters of HIV in Asia, stigma associated with HIV has attracted research attention since the late 1980s. A significant amount of research and resources were invested in documenting the types and frequency of stigma events and their negative impacts, as well as in policy programming to address the stigma against PLWH and their families, especially through mass education providing basic HIV information. Three decades later, however, stigma remains rampant in Thai society, although stigma decreased to some extent after the introduction of ART in early 2000. A recent study drawing on a representative sample of 10,522 adults across Thailand shows that nearly 60% of the population meet the criteria for discriminatory attitudes toward PLWH based on the UNAIDS global indicator. More specifically, close to 70% of the respondents agree that PLWH suffer from stigma and the participants anticipate discriminatory events to happen, close to 60% report a fear of HIV infection when in contact with PLWH, and close to 40% indicate the participants would feel ashamed if they tested positive. In healthcare settings, more than 80% of the staff members are found to have negative attitudes toward PLWH. As a result, PLWH across genders, sexualities, age cohorts, and ethnic groups still report experiences of stigma in their daily lives, as well as constant fear and anxiety for possible repercussions once their serostatus is divulged, leading to suboptimal physical and mental health outcomes. Moreover, those PLWH who belong to marginalized groups, such as transgender women, attribute their suffering to their own personal characteristics and behaviors, rather than to the unjust social institutions, prejudices of mainstream society, and cultural norms of Thailand. A key contributing factor for this slow progress is that the existing interventions often fail to consider the fact that "both stigma and discrimination are deeply rooted in local culture values and follow 'fault lines' in communities", as concluded by Graham Fordham, a medical anthropologist who has conducted ethnographical HIV research in Thailand since the 1990s and extensively reviewed the results of Thai HIV studies published before 2010. Fordham advocated that for stigma reduction interventions to be efficacious, studies need to obtain a "deeper understanding of the culturally specific knowledge used in the generation of stigma and discrimination, as well as a deeper appreciation of the cultural meanings of its concomitants such as isolation and loneliness." As such, this study will emphasize the role of Thai culture, more specifically Buddhist culture, when addressing the stigma and suffering experienced by Thai PLWH.

Buddhist Understanding of HIV Stigma in Thai Culture:

Culture in Thailand is heavily influenced by Buddhism. Similar to other countries in Southeast Asia, Buddhism laid the foundation of Thai culture before the formation of the modern Siamese-Thai state. Buddhism, in particular Theravada Buddhism, as an encompassing ideology and civic religion, has provided a unified, underlying symbolic system for people in Thailand to interpret and organize their day-to-day lives. Indeed, it is estimated that 94% of the Thai population identifies themselves as Buddhists, and nearly all domains of social life have been shaped by Buddhist worldviews.

As influenced by Buddhist concepts of karma, it is thought that poor choices of health include not recognizing and letting go of strong feelings (vedana), which engender craving for, and attachment to, certain drsti (ideas, e.g., stigma and status) or kama (things, e.g., addicting substances), resulting in a sense of dukkha (suffering). To liberate themselves from suffering, individuals are advised to develop insights into the transient nature of the material world, including their "face," or status, and to practice the Noble Fivefold Path (makka), which includes meditation and mindfulness, in hope of reaching a state of enlightenment. Women, as well as members of gender and sexual minorities, are particularly encouraged to practice to grow their spirituality. During the process, individuals become less attached to those strong desires and grow in compassion and acceptance toward themselves and others. Meanwhile, doing actions to accumulate merit, such as practicing good self-management and providing support for others in need, may also help to reduce bad karma and suffering in future lives. As such, within Buddhist culture, the goal of HIV reduction interventions may be assisting PLWH in finding peace and harmony within themselves by gradually "letting go" of those strong desires for status that contribute to their suffering from HIV stigma. Although Buddhist influences in PLWH's experiences and reactions to stigma have been documented in countries such as Thailand and Cambodia, the existing literature focuses on how karma beliefs deter PLWH from seeking help. This study, by contrast, treats Buddhist philosophy as a part of the culture's resources in this regard and seeks to leverage these cultural factors to promote PLWH's coping and resilience.

Conceptualizing Influences of Buddhism on HIV Stigma Among Thai PLWH:

To further contextualize this study, the investigators propose a working conceptual model adapted from a cognitive-behavioral therapy (CBT) model of stigma (the Threat Identification Model) to situate the HIV stigma experienced by PLWH within the social and cultural environment of Thailand. This model highlights how Buddhist philosophy and practice may influence the universal cognitive-behavioral process of HIV stigma. Negative interpretations or attributions of events to one's HIV status reinforces negative attitudes toward oneself, or internal stigma. PLWH also experience elevated physical or emotional reactions as a response to external adverse events or negative attributions and interpretations of those events. These physical or emotional reactions can further reinforce negative appraisals about themselves. The internal stigma can then, in turn, interfere with the self-care engagement of PLWH, although care engagement could also be directly shaped by the external stigma, such as discrimination. Within this framework, the notion of nonattachment to transient social status also alters the results of cognitive appraisals of the stigma and decreases the threat to PLWH themselves. Meditation and mindfulness practices promote PLWH's awareness of changes to physical and emotional states and assists in better managing these reactions. The growing self-compassion and acceptance that can result due to Buddhist practices also help PLWH revise negative attitudes due to HIV status and may serve as better motivation to engage in care.

Adaptation of an Evidence-Based Stigma Reduction Intervention:

To achieve the investigator's goal of developing a tailored stigma reduction intervention, the investigators will adapt the intervention developed by Bogart and colleagues by integrating Buddhist teachings and other Myanmar sociocultural factors into it. The investigators selected Bogart and colleagues' intervention because of the optimal match of its underlying CBT theoretical model to the project's goals.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* self-identify as a Person Living with HIV
* physically well enough to attend counseling sessions and follow-up visits

Exclusion Criteria:

* have a significant condition, such as neurological or cardiovascular diseases, that prevents them from fully participating the study
* unable to communicate
* unable to provide informed consent to participate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Stigma change | weeks 1,4,7,10
  Personalized Stigma and Negative Image subscales of the HIV Stigma Scale Outcome will be used to assess stigma levels. The instrument contains 40-item in totally to measure the stigma perceived by people with HIV to address the respondent's actual experiences or feelings related to having HIV, as well as how other's responses to their HIV status. Subcategories of the scale include personalized stigma subscale, disclosure subscale, negative self-image subscale, and public attitudes subscale. Each stigma item uses a 4-point Likert-type scale (strongly disagree, disagree, agree and strongly agree), with higher values indicating greater agreement with the item.

SECONDARY OUTCOMES:
Care Engagement change | weeks 1,4,7,10
  Patient Activation Measure will be used to assess degree of care engagement. The HCP is a 13-item scale in which clients rate the nature of their interactions with their health care providers on a four-point scale with 1=always true and 4=never. A low score indicates greater provider engagement. The scale was submitted to principal components factor analysis with Varimax rotation. A one-factor solution emerged with an Eigenvalue of 8.6 and explaining 66.5% of the variance. Cronbach's alpha reliability estimate was 0.96.
Buddhism change | weeks 1,4,7,10
  Buddhist COPE Scale will be used to evaluated nonattachment and four immeasurable scales which can determine the level of Buddhist influence in their lives. We included all eight meditation items given to the Buddhist experts-two items described meditation as a Buddhist activity, three concerned meditations as emotion-focused coping, and three assessed problem-focused coping. Four items described equanimity as attempting to find balance in life, and two items focused on equanimity as a major change in lifestyle. Overall, the BCOPE scale used in the present study contained 74 items, with at least eight of the 10 Buddhist experts correctly identifying the scale to which each item belonged. Validation of a Buddhist Coping Measure Among Primarily Non-Asian Buddhists in the United States.
Mindfulness change | weeks 1,4,7,10
  Mindfulness Scale Revised will measure PLWH's practice of mindfulness.
  Mindfulness was measured by the Cognitive and Affective Mindfulness Scale-Revised- Myanmar version (CAMS-R-M), which was translated and adapted from the English version of CAMS-R (Feldman et al. 2007). The 9-item CAMS-R-M included three factors, an Attention factor (e.g., "It is easy for me to concentrate on what I am doing"), Awareness factor (e.g., "I can usually describe how I feel at the moment in considerable detail"), and Acceptance factor (e.g., "I am able to accept the thoughts and feelings I have"). All the items were rated using a 4-point Likert scale (1 = Rarely/Not at all to 4 = Almost Always), with higher total scores reflecting greater mindfulness qualities. In this study, the Cronbach's alpha of the total scale was 0.87, and three-factor structure of CAMS-R-M has been validated by confirmatory factor analysis among PWH (Huang et al., 2021).

CONTACTS AND LOCATIONS:
Locations (1):
- Sanpatong Hospital, Chiang Mai, Thailand